CLINICAL TRIAL: NCT03141983
Title: Anti-Cytokine Therapy for Hemodialysis InflammatION (ACTION): A Phase II Multi-center Study to Evaluate the Safety and Tolerability of Anakinra, an IL-1 Receptor Antagonist, for Patients Treated With Maintenance Hemodialysis
Brief Title: Anti-Cytokine Therapy for Hemodialysis InflammatION
Acronym: ACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 826900; U01DK099919 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-05-05 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: End-Stage Renal Disease
Keywords: ESRD; End-Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra (Active Comparator): Anakinra (Kineret®) is a therapeutic agent that blocks the effects of IL-1 alpha and IL-1 beta by competitively binding to the interleukin-1 type I receptor (IL-1RI). Anakinra is a recombinant, non-glycosylated form of the naturally occurring human interleukin-1 receptor antagonist (IL-1Ra).
  Anakinra will be supplied in pre-filled syringes as a sterile, clear, colorless-to-white, preservative free solution. Each syringe will contain 100 mg in 0.67 ml solution (pH 6.5) containing disodium EDTA (0.12 mg), sodium chloride (5.48 mg), sodium citrate (1.29 mg), and polysorbate 80 (0.70 mg) in Water for Injection, USP.
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Saline (0.9%) will be used as the placebo, supplied in pre-filled syringes as a sterile, clear, colorless-to-white, preservative free solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Anakinra (Kineret®) is a therapeutic agent that blocks the effects of IL-1α and IL-1β by competitively binding to the interleukin-1 type I receptor (IL-1RI). It is a recombinant, non-glycosylated form of the naturally occurring human interleukin-1 receptor antagonist (IL-1Ra) but differs from human IL-1Ra in that it has the addition of a single methionine residue at the amino terminus. It is supplied commercially in single use 1 ml prefilled glass syringes as a sterile, clear, colorless-to-white, preservative free solution. Each syringe contains: 0.67 ml (100 mg) of anakinra in a solution (pH 6.5) containing sodium citrate (1.29 mg), sodium chloride (5.48 mg), disodium EDTA (0.12 mg) and polysorbate 80 (0.70 mg) in Water for Injection, USP.
  Other Names: Kineret®
  Arms: Anakinra
Drug: Placebo — Saline (0.9%) will be used as the placebo, in single use 1 ml prefilled glass syringes as a sterile, clear, colorless-to-white, preservative free solution.
  Arms: Placebo

SUMMARY:
Anti-Cytokine Therapy for Hemodialysis InflammatION (ACTION) is a phase II multi-center study to evaluate the safety and tolerability of anakinra, an IL-1 receptor antagonist, for patients treated with maintenance hemodialysis.

DETAILED DESCRIPTION:
The ACTION Trial will enroll 80 participants being treated with maintenance hemodialysis for end-stage renal disease. Participants will be randomized to receive Anakinra, 100 mg administered intravenously 3 times per week at the end of the hemodialysis session, or matched placebo. The duration of study drug administration is 24 weeks. There will be an additional 24 weeks of follow-up after study drug administration has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Maintenance hemodialysis therapy 3 times per week for end-stage renal disease
2. ≥6 months since hemodialysis initiation
3. C-reactive protein measured by high sensitivity assay (hsCRP) ≥2.0 mg/L at screening and within 10 days prior to randomization
4. Most recent single pool Kt/V > or = 1.2 within 30 days prior to first screening visit
5. Negative tuberculosis interferon gamma release assay (e.g. Quantiferon-TB Gold) for tuberculosis unless documented treatment for a) positive PPD, b) positive interferon gamma release assay, or c) tuberculosis.
6. Negative human immunodeficiency virus (HIV) antibody test, negative hepatitis C Ab test unless viral clearance following direct antiviral therapy is documented, and negative hepatitis B surface antigen positivity.
7. For women of childbearing potential, willingness to use a highly effective method of birth control for up to 4 weeks after the last dose of anakinra.
8. Ability to provide informed consent

Exclusion Criteria:

1. Current or anticipated use of a hemodialysis central venous catheter
2. Acute bacterial infection, including vascular access infection, within 60 days prior to screening unless treated with antibiotics and resolved. Any chronic bacterial infection (e.g., osteomyelitis or bronchiectasis)
3. Hospitalization within 30 days unless for vascular access procedure
4. Cirrhosis
5. Malignancy within the past 5 years with exception of basal or squamous cell carcinoma
6. Use of an immunosuppressive drug within the past 3 months except low doses of oral corticosteroids (total daily dose ≤10 mg/day of prednisone or equivalent)
7. Receipt of live vaccine within the past 3 months. Live vaccines include Varicella zoster, measles, oral polio, rotavirus, yellow fever, and the nasal spray influenza vaccine
8. Absolute neutrophil count (ANC) <2,500 cells/mm3 (2.5 x 109 cells/L)
9. Platelet count <100,000/mm3 (100 x 109/L)
10. Known allergy to anakinra
11. Anticipated kidney transplantation, change to peritoneal dialysis, or transfer to another dialysis unit within 9 months
12. Expected survival less than 9 months
13. Pregnancy, anticipated pregnancy, or breastfeeding
14. Incarceration
15. Receipt of an investigational drug within the past 30 days
16. Current or anticipated participation in another intervention study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dember, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - The George Washington University, Washington D.C., District of Columbia
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington Kidney Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Research results will be made available to the scientific community and public in a timely manner. The primary method by which data will be shared with the scientific community will be through peer-reviewed publications and presentation at scientific and professional society meetings. In addition, data and results will be submitted to the NIH in the annual progress reports required under the terms and conditions of the funding award. This study will also be registered with clinicaltrials.gov before initiation.
  Data from the study will be submitted to the NIDDK Data Repository in accordance with the NIDDK Data Sharing policy. The policy requires that data sets be transferred no later than 2 years after study completion or 1 year after publication of the primary results, whichever comes first. Through the repository, the study data will be made available to external investigators.

RESULTS

PARTICIPANT FLOW:
Groups:
- Anakinra: Anakinra (Kineret®) is a therapeutic agent that blocks the effects of IL-1 alpha and IL-1 beta by competitively binding to the interleukin-1 type I receptor (IL-1RI). Anakinra is a recombinant, non-glycosylated form of the naturally occurring human interleukin-1 receptor antagonist (IL-1Ra).
  Anakinra will be supplied in pre-filled syringes as a sterile, clear, colorless-to-white, preservative free solution. Each syringe will contain 100 mg in 0.67 ml solution (pH 6.5) containing disodium EDTA (0.12 mg), sodium chloride (5.48 mg), sodium citrate (1.29 mg), and polysorbate 80 (0.70 mg) in Water for Injection, USP.
  Anakinra: Anakinra (Kineret®) is a therapeutic agent that blocks the effects of IL-1α and IL-1β by competitively binding to the interleukin-1 type I receptor (IL-1RI). It is a recombinant, non-glycosylated form of the naturally occurring human interleukin-1 receptor antagonist (IL-1Ra) but differs from human IL-1Ra in that it has the addition of a single methionine residue at the amino terminus. It is supplied commercially in single use 1 ml prefilled glass syringes as a sterile, clear, colorless-to-white, preservative free solution. Each syringe contains: 0.67 ml (100 mg) of anakinra in a solution (pH 6.5) containing sodium citrate (1.29 mg), sodium chloride (5.48 mg), disodium EDTA (0.12 mg) and polysorbate 80 (0.70 mg) in Water for Injection, USP.
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 38 | 42
Completed | 30 | 34
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Placebo | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.0) | 54.1 (13.5) | 56.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 33 | 39 | 72
  Unknown or Not Reported | 0 | 0 | 0
hsCRP, mg/L [Median (Inter-Quartile Range); unit: mg/L] | 7.2 [5.4 to 15.8] | 7.2 [5.8 to 16.0] | 7.2 [5.8 to 16.0]

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Anakinra, for Patients Receiving Maintenance Hemodialysis
Description: The primary safety endpoint is serious adverse events per patient-year.
Time Frame: 48 Weeks (after the 24-week treatment period and the 24-week post-treatment period)
Measure: Number; unit: events per patient-year
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
events per patient-year | 2.71 | 2.74

2. Primary Outcome: Change in Log-transformed Circulating CRP Concentration After 24 Weeks of Treatment for Patients Receiving Maintenance Hemodialysis
Description: For this outcome, CRP measurements from Baseline and Week 24 were compared.
Time Frame: Change from Baseline to 24 Weeks (end of treatment phase)
Measure: Mean (Standard Deviation); unit: Log (mg/L)
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
Log (mg/L) | -0.4 (0.9) | -0.2 (0.7)

3. Secondary Outcome: Number of Participants With Adverse Events That Preclude Further Treatment With the Study Agent
Description: Adverse events were one measure used to assess safety and tolerability of anakinra, for patients receiving maintenance hemodialysis. This measure assessed the number of participants with adverse events that precluded further treatment with the study agent.
Time Frame: 24-week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
Participants | 3 | 1

4. Secondary Outcome: Safety and Tolerability of Anakinra, for Patients Receiving Maintenance Hemodialysis - Infections
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
Participants | 5 | 11

5. Secondary Outcome: Safety and Tolerability of Anakinra, for Patients Receiving Maintenance Hemodialysis - Neutropenia
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
Participants | 1 | 0

6. Secondary Outcome: Safety and Tolerability of Anakinra, for Patients Receiving Maintenance Hemodialysis - Thrombocytopenia
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
Participants | 0 | 0

7. Secondary Outcome: Safety and Tolerability of Anakinra, for Patients Receiving Maintenance Hemodialysis - Systemic Hypersensitivity Reactions
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
Participants | 1 | 0

8. Secondary Outcome: Change in Markers of Inflammation and Oxidative Stress - IL-1β pg/ml
Description: Change in circulating markers of inflammation and oxidative stress between baseline and end of treatment
Time Frame: change after 24 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
pg/ml | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.0]

9. Secondary Outcome: Change in Markers of Inflammation and Oxidative Stress - IL-6, pg/mL
Time Frame: change after 24 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
pg/mL | -0.7 [-2.4 to -0.3] | 0.0 [-1.0 to 0.7]

10. Secondary Outcome: Change in Markers of Inflammation and Oxidative Stress - IL-10, pg/mL
Time Frame: change after 24 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
pg/mL | 0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1]

11. Secondary Outcome: Change in Markers of Inflammation and Oxidative Stress - TNF Alpha, pg/ml
Time Frame: change after 24 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
pg/ml | -0.2 [-1.0 to 0.1] | 0.0 [-0.3 to 0.7]

12. Secondary Outcome: Change in Markers of Inflammation and Oxidative Stress - Albumin, g/dL
Time Frame: change after 24 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
g/dL | 0.0 [-0.2 to 0.1] | 0.0 [-0.2 to 0.2]

13. Secondary Outcome: Change in Patient-reported Indicators of Fatigue After 24 Weeks of Treatment
Description: Change in patient reported outcomes using the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue scale from Baseline to Week 24.
  To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
  All participants were assessed with the same scoring system.
Time Frame: 24 Weeks (end of treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
score on a scale | -4.9 (12.1) | -0.4 (8.7)

14. Secondary Outcome: Change in Patient-reported Indicators of Depression After 24 Weeks of Treatment for Patients Receiving Maintenance Hemodialysis
Description: Change in patient reported outcomes using the Beck Depression Inventory - II (BDI-II) scale at baseline, Weeks 12, 24 and 28.
  The instrument uses a 21-item self-report inventory measuring the severity of depression in adolescents and adults.The standard cut-offs are as follows: 0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
Time Frame: 24 Weeks (end of treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
score on a scale | -0.9 (5.7) | -0.1 (7.5)

15. Secondary Outcome: Change in Burden of Patient-reported Symptoms After 24 Weeks of Treatment for Patients Receiving Maintenance Hemodialysis
Description: Mean change in patient reported outcomes using the Dialysis Symptom Index, Burden subscale
  The DSI is a 30-question instrument assessing whether participants report a particular symptom during the past week and the severity of that symptom. Symptom burden is assessed using 30 "yes/no" questions. The scale is a count of the number of "yes" responses. The minimum is 0. The maximum is 30. The mean change in score after 24 weeks of treatment was measured. A lower score is better as a higher score indicates greater symptom burden.
Time Frame: Change after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
score on a scale | 0.2 (5.6) | 0.3 (3.8)

16. Secondary Outcome: Change in Severity of Patient-reported Symptoms After 24 Weeks of Treatment for Patients Receiving Maintenance Hemodialysis
Description: Change in patient reported outcomes using the Dialysis Symptom Index, Severity subscale
  The DSI severity subscale includes 30-questions assessing whether a symptom is present (previous outcome - burden subscale). The severity of each symptom that was reported as being present was assessed by asking patients to rate the degree to which the symptom was bothersome using a five-point Likert scale (1 = "not at all bothersome" to 5 = "bothers very much"). Higher scores indicating greater symptom severity. The minimum score is 30, the maximum score is 150. The mean change was used to measure this outcome.
Time Frame: Change after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
score on a scale | -4.0 (24.4) | -0.3 (15.1)

17. Secondary Outcome: Change in Patient-reported Indicators of Quality of Life After 24 Weeks of Treatment for Patients Receiving Maintenance Hemodialysis
Description: Change in patient reported outcomes using the Kidney Disease - Quality of Life subscale of the SF-12 (KDQOL SF-12) at baseline, Weeks 12, 24 and 28.
  A higher score reflects a more favorable health state. The questionnaire consists of 24 questions and the total possible score sum is 0-100. Items in the same scale are averaged to create scale scores.
Time Frame: 24 Weeks (end of treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
score on a scale | -3.5 (21.5) | -3.3 (14.2)

18. Secondary Outcome: Change in Measure of Muscle Strength (Hand Grip Strength) After 24 Weeks of Treatment for Patients Receiving Maintenance Hemodialysis
Description: Change in measurement of hand grip strength using a standard dynamometer at baseline, Weeks 12, 24 and 28. This was measured in kg using the dominant hand.
Time Frame: 24 Weeks (end of treatment phase)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 38 | 42
kilograms | -0.5 (4.1) | -0.4 (3.9)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | Anakinra | Placebo
All-Cause Mortality (participants affected / at risk) | 2/38 | 4/42
Serious Adverse Events (participants affected / at risk) | 17/38 | 23/42
Other Adverse Events (participants affected / at risk) | 7/38 | 11/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=38) | Placebo (N=42)
hypotension (Vascular disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Vascular Access Complication (Vascular disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Kidney transplant (Surgical and medical procedures) | 1 | 1
Severe central canal stenosis (Nervous system disorders) | 1 | 0
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Clotted AVF (Vascular disorders) | 0 | 3
Thrombolysis (Vascular disorders) | 0 | 1
Sudden cardiac death (Cardiac disorders) | 0 | 1
Epiretinal membrane (Eye disorders) | 0 | 1
non-ST elevated myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac catheterization (Cardiac disorders) | 0 | 1
acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
autonomic dysfunction (Nervous system disorders) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 2
hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Norovirus associated gastroenteritis (Gastrointestinal disorders) | 0 | 1
COVID19 (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=38) | Placebo (N=42)
Sinusitis (Infections and infestations) | 1 | 0
COVID (Infections and infestations) | 1 | 1
neutropenia (Blood and lymphatic system disorders) | 1 | 0
Flu (Infections and infestations) | 1 | 1
Urticaria (Immune system disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Acute osteomyelitis of left foot (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Norovirus (Infections and infestations) | 0 | 1
Non-serious infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Pyelonephritis of transplanted kidney (Infections and infestations) | 0 | 1
Toe blisters (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03141983/Prot_SAP_000.pdf